CLINICAL TRIAL: NCT05917236
Title: Biliary Atresia and Preduodenal Portal Vein
Brief Title: Biliary Atresia With Rare Associations, a Case Report
Acronym: BA
Status: Completed | Type: Observational
Sponsor: Sarah Magdy Abdelmohsen (Other)
Responsible Party: Sponsor-Investigator, Sarah Magdy Abdelmohsen, Principal Investigator, Aswan University Hospital
Organization: Aswan University Hospital (Other)
Other Study IDs: AswanUH4
Record Dates: First submitted 2022-10-26; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: BA - Biliary Atresia
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: hepato-portoentostomy — the retro-colic Roux-en-Y limb of the jejunum, and finally hepato-portoentostomy (Kasai operation)
  Other Names: (Kasai operation)

SUMMARY:
Background: It is not often written in medical journals that preduodenal portal vein, biliary atresia, intestinal malrotation, and situs inversus totalis are all related.

Case reports: A two-month-old female infant had biliary atresia type III, situs inversus totalis, midgut malrotation, and preduodenal portal vein. She had been operated on by the Kasai procedure (hepato-portoenterostomy).

Discussion: It is important to carefully look into the relationship between preduodenal portal vein and biliary atresia because the patient at a risk of injury from this aberrant vein at operative intervention.

DETAILED DESCRIPTION:
A full-term female infant, G1P1, weighing 3450 g at birth, was referred to our department at the age of 2 months old with severe jaundice and poor feeding. The mother reported yellow sclera and skin, lightning-colored stool, and dark colored urine a few days after birth, which were progressively aggravated.

On physical examination, the infant had an olive-green colored sclera and skin with an itching mark, a pale clay stool in the diaper, a law grade fever of 37.8°C, a weight of 3870 g, a pulse rate of 138 b/m, and a respiratory rate of 38 b/m. The heart sounds and breath sounds were normal. The abdomen was soft and lax on examination. The liver was two fingers below the costal margin. The intestinal sound was normal.

The laboratory investigation revealed that total bilirubin was elevated at 7 mg/dl, direct bilirubin was elevated at 4 mg/dl, GGT was elevated at 157,1 U/L, alkaline phosphatase was elevated at 279 U/L, and albumin was decreased at 3.4 g/dL.

Abdominal ultrasonography revealed a triangular cord sign in the liver hilum, an absent gall bladder, and a normal-sized spleen on the right side behind the liver. A chest x-ray revealed dextrocardia. The HIDA scan revealed failure of radioisotope excretion in the duodenum . Non-contrast magnetic resonance cholangiopancreatography (MRCP) showed that the common hepatic duct and the common bile duct could not be seen. Preoperative percutaneous liver biopsy reported liver fibrosis, bile ductules proliferation and cholestasis.

An experienced pediatric surgeon obtained the decision for exploratory laparotomy by right subcostal abdominal incision. The spleen is located in the right upper quadrant behind the liver. Extracorporealization of the liver is done . The gall bladder was rudimentary. On further exploration, the principle investigator also found intestinal malrotation (IM) and PDPV. All extrahepatic bile ducts were absent; type III portal atresia. The portal palate was dissected easily and the rudimentary gall bladder was removed.

Widening of the narrow base of the intestinal mesentery, then reconstruction of the retro-colic Roux-en-Y limb of the jejunum, and finally hepato-portoentostomy (Kasai operation) was done . A wedge liver biopsy obtained reported ductular proliferation, hepatic fibrosis, and bile plugs; a feature suggestive of biliary obstruction.

The post-operative follow-up of the patient revealed features of bile drainage in the intestine; the stool returned to its normal brawn color; and the yellow skin color was slightly improved. Total bilirubin was 4 mg/dl and direct bilirubin was 2 mg/dl. The patient was discharged on the tenth post-operative day.

ELIGIBILITY:
Inclusion Criteria:

- Biliary atresia with another syndrome

Exclusion Criteria:

* Biliary atresia alone

Ages: 2 Months to 3 Months | Sex: Female
Age Groups: Child
Study Population: one case reports
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Is the infant will still a live or he will dies? | from 3 weeks to one year follow up
  Is the infant will continue his life up to one year or he will dies during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Abdelmohsen, Lecturer, Study Director — Aswan University Hospital
Locations (1):
- Aswan university, Aswān, Sahary, Egypt

IPD SHARING:
Plan to Share IPD: Undecided